CLINICAL TRIAL: NCT05697809
Title: A Multi-Center, Randomized, Parallel-Group, Phase 2, Masked, Three-Arm Trial to Compare Safety, Tolerability, Efficacy, and Durability of Two Dose Levels of Suprachoroidal Sustained-Release OXU-001 (Dexamethasone Microspheres; DEXAspheres®) Using the Oxulumis® Illuminated Microcatheterization Device Compared With Intravitreal Dexamethasone Implant (OZURDEX®) in Subjects With Diabetic Macular Edema (OXEYE)
Brief Title: Suprachoroidal Sustained-Release OXU-001 Compared to Intravitreal Ozurdex® in the Treatment of Diabetic Macular Edema
Acronym: OXEYE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxular Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OXUCT-102 - OXEYE
Record Dates: First submitted 2023-01-13; First posted 2023-01-26 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Macular Edema
Keywords: Macular Edema; Edema; Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; Anti-Inflammatory Agents; Glucocorticoids; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Physiological Effects of Drugs; Immunosuppressive Agents; Immunologic Factors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Dexamethasone; Suprachoroidal Microcatheterization; Illuminated Microcatheterization; Sustained-Release
MeSH Terms: conditions — Macular Edema; Edema; Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases

STUDY DESIGN:
Intervention Model Description: The trial was designed to include previously IVT anti-VEGF treated (in Part A and B) and treatment-naive (in Part B only) DME subjects.
  In Part A, approximately 18 subjects will be randomly assigned (ratio 1:1) to receive either a mid-dose or high-dose of suprachoroidal OXU-001.
  In Part B, approximately 110 subjects will be randomly assigned (ratio 2:2:1) to receive a single treatment of either suprachoroidal OXU-001 Dose 1, or Dose 2 or intravitreal Ozurdex® Note: Due to a non-safety related sponsor decision in Dec 2024 trial recruitment was stopped after only 3 subjects randomized and treated in Part A of the clinical trial. Part B was therefore not initiated.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A is open-label, no masking. Part B is masked for the subject and the outcomes assessing site team and central reading center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- A1: OXU-001 / Mid dose (Experimental): The Oxulumis® device will be used for the administration of OXU-001 (sustained release dexamethasone acetate) via suprachoroidal microcatheterization. A single treatment with dose level 1 (mid dose) will be applied.
  Interventions: Drug: OXU-001; Device: Semi-automated suprachoroidal illuminated microcatheter
- A2: OXU-001 / High Dose (Experimental): The Oxulumis® device will be used for the administration of OXU-001 (sustained release dexamethasone acetate) via suprachoroidal microcatheterization. A single treatment with dose level 2 (high dose) will be applied.
  Interventions: Drug: OXU-001; Device: Semi-automated suprachoroidal illuminated microcatheter
- B1: OXU-001 / Mid Dose (Experimental): The Oxulumis® device will be used for the administration of OXU-001 (sustained release dexamethasone acetate) via suprachoroidal microcatheterization. A single treatment with dose level 1 (mid dose) will be applied.
  Interventions: Drug: OXU-001; Device: Semi-automated suprachoroidal illuminated microcatheter
- B2: OXU-001 / High Dose (Experimental): The Oxulumis® device will be used for the administration of OXU-001 (sustained release dexamethasone acetate) via suprachoroidal microcatheterization. A single treatment with dose level 2 (high dose) will be applied. This dose may be adpated based on the outcome of a Week 6 data review of Part A
  Interventions: Drug: OXU-001; Device: Semi-automated suprachoroidal illuminated microcatheter
- B3: Ozurdex® (Active Comparator): A single treatment with intravitreal Ozurdex®
  Interventions: Drug: Ozurdex® Ophthalmic Intravitreal Implant

INTERVENTIONS:
Drug: OXU-001 — Suprachoroidal sustained release dexamethasone acetate
  Other Names: DEXAspheres®
  Arms: A1: OXU-001 / Mid dose; A2: OXU-001 / High Dose; B1: OXU-001 / Mid Dose; B2: OXU-001 / High Dose
Device: Semi-automated suprachoroidal illuminated microcatheter — Ophthalmic administration device
  Other Names: Oxulumis®
  Arms: A1: OXU-001 / Mid dose; A2: OXU-001 / High Dose; B1: OXU-001 / Mid Dose; B2: OXU-001 / High Dose
Drug: Ozurdex® Ophthalmic Intravitreal Implant — Ophthalmic dexamethasone intravitreal implant
  Other Names: intravitreal dexamethasone implant
  Arms: B3: Ozurdex®

SUMMARY:
The purpose of this clinical trial is to compare safety, tolerability, efficacy, and durability of two dose levels of suprachoroidal sustained-release OXU-001 (dexamethasone microspheres; DEXAspheres®) using the Oxulumis® illuminated microcatheterization device compared with intravitreal dexamethasone implant (OZURDEX®) in subjects with diabetic macular edema.

DETAILED DESCRIPTION:
Fifty-two (52) week phase 2 trial with two parts. Part A is an open-label, randomized, single-dose two treatment arm comparison of two dose levels of sustained-release suprachoroidal OXU-001 (DEXAspheres® administered using the Oxulumis® illuminated microcatheterization device) in subjects with Diabetic Macular Edema.

--- Part A was only partially recruited due a non-safety related sponsor decision to stop further recruitment after 3 randomized and treated subjects.

--- Part B is a randomized, masked, active comparator, single-dose, three treatment arm comparison of two dose levels of suprachoroidal OXU-001 and IVT Ozurdex® to evaluate the safety, tolerability, efficacy, and durability in subjects with Diabetic Macular Edema (DME).

--- Part B was not initiated due a non-safety related sponsor decision in Dec 2023.

--- In Part A, after a screening period, approximately 18 adult female or male subjects will be randomized in a 1:1 ratio to receive a single administration of one of two dose levels of OXU-001 (mid-dose or high-dose).

In Part B, after a screening period, approximately 110 adult female or male subjects will be randomized in a 2:2:1 ratio to receive a single administration of one of two dose levels of OXU-001 (Dose 1 or Dose 2) or Ozurdex®.

From Week 12, subjects will be assessed for the need for follow-on treatment. The follow-up period after treatment administration will be up to fifty-two (52) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* Diabetic Macular edema involving the center of the fovea in the study eye
* Best corrected visual acuity in the study eye between 34 and 78 (early treatment of diabetic retinopathy study) ETDRS letters

Exclusion Criteria:

* Macular edema is considered due to a cause other than diabetes mellitus in the study eye
* Condition, in the study eye, in which visual acuity is not expected to improve from the resolution of macular edema
* Macular laser photocoagulation or panretinal laser photocoagulation in the study eye performed within 16 weeks prior to screening
* Active proliferative diabetic retinopathy (PDR) or sequelae of PDR in the study eye
* Prior treatment with anti-VEGF in the study eye:

  1. Treatment naïve group (Part B), any IVT anti-VEGF treatments in the study eye are exclusionary regardless of the time interval since injection.
  2. Previously treated group (Part A and B), subjects in the previously treated group are excluded if they meet any of the below criteria for the study eye at screening:

     1. Subject has received less than 3 anti-VEGF injections since treatment initiation (at least three injections must have been received for eligibility).
     2. Time interval between the first anti-VEGF injection and screening is more than 40 weeks.
     3. Last injection with ranibizumab or bevacizumab within 4 weeks prior to screening.
     4. Last injection with aflibercept within 8 weeks prior to screening.
     5. Last injection with faricimab or brolucizumab within 12 weeks prior to screening.
     6. Prior treatment with SUSVIMO (Port Delivery System) implant is exclusionary.
* Prior ocular treatment with steroid injections (periocular, subtenon, intravitreal) or intravitreal implants in the study eye.
* Prior treatment with suprachoroidal steroids in the study eye is exclusionary.
* Active malignancy or history of malignancy within the past 5 years
* Uncontrolled diabetes with a hemoglobin A1c (HbA1c) more than 12% or any other uncontrolled systemic disease at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Asmus, MD, Study Director — Oxular Limited
Locations (9):
- United States (8):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Blue Ocean Clinical Research West, Clearwater, Florida
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Retina Consultants of Minnesota, Minneapolis, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Retina Consultants of Texas, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Retinal Consultants of Texas - San Antonio, San Antonio, Texas
- Emmanuelli Research and Development Center, LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose | B1: OXU-001 / Mid Dose | B2: OXU-001 / High Dose | B3: Ozurdex®
Started | 1 | 2 | 0 | 0 | 0
Completed | 1 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 | 55.5 (2.1) | 58.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 1 | 2 | 3
Best-Corrected Visual Acuity (BCVA) - Study EYE [Mean (Standard Deviation); unit: letters read correctly on ETDRS charts] | 61.0 | 64.0 (9.9) | 63.0 (7.2)
Central Subfield Thickness (Study Eye) [Mean (Standard Deviation); unit: µm] — assessed at the Baseline Visit before treatment
  µm | 417.0 | 502.5 (7.8) | 474.0 (49.7)

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Ocular and Systemic Treatment Emergent Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest
Description: Treatment-emergent adverse events are defined as events emerging following administration of study treatment (OXU-001 administered with the Oxulumis suprachoroidal administration device) at Visit 2 (Baseline, Day 0)
Time Frame: Day 0 up to Week 52
Population: Safety Analysis Set - - Number of Participants with at least 1 event
Measure: Count of Participants; unit: Participants
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
Number analyzed (Participants) | 1 | 2
Participants
  Number of Participants with Ocular Treatment Emergent Adverse Events | 0 | 2
  Number of Participants with Systemic (Non-Ocular) Treatment Emergent Adverse Events | 1 | 2
  Number of Participants with Ocular Serious Adverse Events | 0 | 0
  Number of Participants with Systemic (Non-Ocular) Serious Adverse Events | 0 | 0
  Number of Participants with Adverse Events of Special Interest | 0 | 0

2. Primary Outcome: Frequency and Severity of Treatment-emergent Adverse Device Effects
Description: Treatment-emergent adverse device effects are defined as effects emerging following administration of study treatment at Visit 2 (Baseline, Day 0)
Time Frame: Day 0 up to Week 52
Population: Safety Analysis Set - - Number of Participants with at least 1 event
Measure: Count of Participants; unit: Participants
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
Number analyzed (Participants) | 1 | 2
Participants
  Number of Participants with Adverse Device Effects | 0 | 0
  Number of Participants with Serious Adverse Device Effects | 0 | 0

3. Other Pre Specified Outcome: Mean Change in Best-Corrected Visual Acuity (BCVA) Compared to Baseline, Visit 2, Day 0
Description: Assessed using the Early Treatment of Diabetic Retinopathy (ETDRS) methodology. All BCVA assessments in the study eye need to be performed in duplicate. The mean of both BCVA assessments was calculated, if both ETDRS letters scores differ by more than 5 letters, the better (higher) ETDRS letter score will be used.
Time Frame: Week 24
Population: Full Analysis Set, Study Eye, Number of Participants with at least 1 post baseline assessment
Measure: Mean (Standard Deviation); unit: letters read correctly on ETDRS charts
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
Number analyzed (Participants) | 1 | 2
letters read correctly on ETDRS charts | 9.0 | 6.5 (0.7)

4. Other Pre Specified Outcome: Mean Change in Best-Corrected Visual Acuity (BCVA) Compared to Baseline, Visit 2, Day 0
Description: as for outcome 3
Time Frame: Week 52
Population: Full Analysis Set, Study Eye
Measure: Mean (Standard Deviation); unit: letters read correctly on ETDRS charts
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
Number analyzed (Participants) | 1 | 2
letters read correctly on ETDRS charts | 11.0 | 10.5 (3.5)

5. Other Pre Specified Outcome: Mean Change in Central Subfield Thickness (CST) Compared to Baseline, Visit 2, Day 0
Description: Assessed using Spectral-Domain Optical Coherence Tomography (SD-OCT) using the Central Subfield Thickness values calculated by the software of the SD-OCT devices allowed in the OXEYE clinical trial.
Time Frame: Week 24
Population: Full Analysis Set, Study Eye
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
Number analyzed (Participants) | 1 | 2
µm | -16.0 | -165.0 (45.3)

6. Other Pre Specified Outcome: Mean Change in Central Subfield Thickness (CST) Compared to Baseline, Visit 2, Day 0
Description: as for outcome 5
Time Frame: Week 52
Population: Full Analysis Set, Study Eye
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
Number analyzed (Participants) | 1 | 2
µm | -10.0 | -81.5 (31.8)

7. Other Pre Specified Outcome: Time Interval to Subjects Requiring follow-on Treatment (From Baseline, Visit 2, Day 0)
Description: Timepoint for meeting pre-specified, protocol-defined criteria of disease activity recurrence. Disease activity was assessed based on Best-Corrected Visual Acuity using the Early Treatment of Diabetic Retinopathy Screening methodology and the central subfield thickness using Spectral-Domain OCT. If criteria were not met throughout Week 52, 365 days were entered.
Time Frame: From Week 12 through Week 52
Population: Full Analysis Set, Study Eye
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
Number analyzed (Participants) | 1 | 2
Days | 365 | 118.5 (6.4)

ADVERSE EVENTS:
Time Frame: Day 0 up to Week 52
Description: Treatment-emergent ocular adverse events are defined as an ocular event that emerges following the start of administration of OXU-001 with the Oxulumis® microcatheter at Visit 2 (Baseline, Day 0)
Arm/Group | A1: OXU-001 / Mid Dose | A2: OXU-001 / High Dose
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1: OXU-001 / Mid Dose (N=1) | A2: OXU-001 / High Dose (N=2)
Conjunctival Hemorrhage (Eye disorders) | 0 (0) | 2 (2) — Study Eye
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Right Humerus Fracture
Worsening of Diabetes Mellitus (Vascular disorders) | 0 (0) | 1 (1)
Worsening of Arterial Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT05697809/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT05697809/SAP_002.pdf